CLINICAL TRIAL: NCT04051736
Title: a Randomized, Controlled Clinical Trial of Immunogenicity and Safety of Sabin-based Inactivated Polio Vaccine Replacing Salk-based Inactivated Polio Vaccine
Brief Title: Immunogenicity and Safety of Sabin-IPV Replacement Vaccination
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: China National Biotec Group Company Limited (Industry)
Collaborators: Beijing Institute of Biological Products Co Ltd. (Industry); Beijing Center for Disease Control and Prevention (Other Government); Peking University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: ChinaNBG
Record Dates: First submitted 2019-08-08; First posted 2019-08-09 (Actual); Last update posted 2020-09-09 (Actual); Status verified 2020-09

CONDITIONS: Vaccination
MeSH Terms: interventions — Poliovirus Vaccine, Inactivated

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- group 1 (Experimental): 180 2-month-old subjects will be enrolled with vaccination schedule as follows: 1st: Salk-IPV; 2nd: Sabin-IPV; 3rd: Sabin-IPV
  Interventions: Biological: Inactivated Polio Vaccine
- group 2 (Active Comparator): 180 2-month-old subjects will be enrolled with vaccination schedule as follows: 1st: Salk-IPV; 2nd: Salk-IPV; 3rd: Salk-IPV
  Interventions: Biological: Inactivated Polio Vaccine

INTERVENTIONS:
Biological: Inactivated Polio Vaccine — Inactivated Polio Vaccine at age of 2,3,4 months old, respectively

SUMMARY:
This study replaced the 2nd and 3rd dose of Salk-IPV (produced by Sanofi) with Sabin-IPV (produced by CNBG) and then reviewed the safety and immunogenicity of the vaccination, aiming to acquire scientific evidence for the feasibility of immunization involving different viral strains replacement.

DETAILED DESCRIPTION:
It is required by China Food and Drug Administration (CFDA) that considering in the real situation IPV receivers may be immuned by different viral strains of this vaccine, a phase 4 clinical trial aiming to demonstrate the safety and immunogenicity of the immunization schedule should be carried out. To be specific, the subjects were divided into 2 groups.

Group 1 received Salk-IPV+Sabin-IPV+Sabin-IPV respectively at the age of 2,3,4 months old.

Group 2 received Salk-IPV+Salk-IPV+Salk-IPV respectively at the age of 2,3,4 months old.

Blood sample was collected before vaccination and 30 days after the third dose of vaccination. Neutralization antibody against type I, Type II and Type III poliomyelitis virus were detected to evaluate the seroprotection rates and antibody geometric mean concentrations. The safety of both immunization schedule will also been monitored.

ELIGIBILITY:
Inclusion Criteria:

* subjects aged from 60 days to 89 days old at the date of recruitment;
* with informed consent signed by parent(s) or guardians;
* parent(s) or guardians are able to attend all planned clinical appointments and obey and follow all study instructions;
* subjects did not receive any vaccines within 14 days;
* axillary temperature ≤37.0℃

Exclusion Criteria:

* allergic to any ingredient of vaccine or with allergy history to any vaccine;
* acute febrile disease or infectious disease;
* serious chronic diseases;
* any other factor that makes the investigator determines the subject is unsuitable for this study;

Ages: 60 Days to 89 Days | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 360 (Actual)
Dates: Start 2018-03-01 (Actual); Primary Completion 2018-12-28 (Actual); Study Completion 2020-08-31 (Actual)

PRIMARY OUTCOMES:
Seroconversion rate | 4 months
  determine the seroconversion rate of both groups

SECONDARY OUTCOMES:
Neutralizing antibody titers | 4 months
  Measure neutralizing antibody titers against poliovirus type I, II and III

OTHER OUTCOMES:
number of participants who experience adverse events | 6 months
  analyse the number and rate of vaccine participants who have adverse events following immunization

CONTACTS AND LOCATIONS:
Overall Officials: Jiang WU, Study Director — Beijing Center for Disease Control and Prevention
Locations (1):
- Beijing Center for Disease Control and Prevention, Beijing, Beijing Municipality, China

REFERENCES:
- [Derived] Chen H, Gao Z, Bai S, Liu X, Han S, Xiao Y, Liu F, Yu Y, Sun H, Yang X. Immunogenicity and safety of sabin-strain based inactivated poliovirus vaccine replacing salk-strain based inactivated poliovirus vaccine: An innovative application of different strain-IPVs replacement. Vaccine. 2021 Apr 22;39(17):2467-2474. doi: 10.1016/j.vaccine.2021.02.073. Epub 2021 Mar 31. PMID 33810904